CLINICAL TRIAL: NCT03867656
Title: Effects of Gut Peptides on Bone Remodeling. KS-4-Diabetes-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Kirsa Skov-Jeppesen, Principal Investigator, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: KS-4-Diabetes-19
Record Dates: First submitted 2019-03-05; First posted 2019-03-08 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Bone resorption; Bone formation; CTX; P1NP; GLP-2; GIP; Bone turnover; Bone remodeling
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Bone Resorption

STUDY DESIGN:
Intervention Model Description: The study is a crossover study with the following interventions: GLP-2, GIP, and placebo.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GLP-2 (Experimental): Glucagon-like peptide 2
  Interventions: Other: GLP-2
- GIP (Experimental): Glucose-dependent insulinotropic polypeptide
  Interventions: Other: GIP
- Placebo (Placebo Comparator): Saline
  Interventions: Other: Placebo

INTERVENTIONS:
Other: GLP-2 — GLP-2 injection
  Arms: GLP-2
Other: GIP — GIP injection
  Arms: GIP
Other: Placebo — Placebo injection
  Arms: Placebo

SUMMARY:
Both GLP-2 and GIP reduce the bone resorption (measured as CTX) in healthy persons. In this study, we will investigate wether GLP-2 and GIP is reducing CTX in persons with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 25 to 70 years old.
* Type 2 diabetes.
* In Metformin or sulfonylureas

Exclusion Criteria:

* Treatment with other antidiabetics
* Osteopososis or gastrointestinal disease
* Smoking
* Long term steroid treatment
* Weight change more than 3 kg within the last 3 months.
* Overweight or intestinal surgery

Ages: 25 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
CTX | -10 minutes to 240 minutes
  Bone resorption measured as collagen type 1 C-terminal telopeptide (CTX) in serum.
P1NP | -10 minutes to 240 minutes
  Bone formation measured as procollagen type 1 N-terminal propeptide (P1NP) in serum.

SECONDARY OUTCOMES:
PTH | -10 minutes to 240 minutes
  PTH measured in serum
Sclerostin | -10 min to 240 min.
  Bone marker.
Glucose | -10 minutes to 240 minutes
  Measured in serum
Insulin | -10 minutes to 240 minutes
  Measured in serum
C-peptide | -10 minutes to 240 minutes
  Measured in serum
GIP | -10 minutes to 240 minutes
  Glucose-dependent insulinotropic polypeptide measured in plasma.
GLP-2 | -10 minutes to 240 minutes
  Glucagon-like peptide 2 measured in plasma.
Glucagon | -10 minutes to 240 minutes
  Glucagon measured in plasma
Blood pressure | -10 minutes to 240 minutes
  Measured before blood sampling
Heart rate | -10 minutes to 240 minutes
  Measured before blood sampling

CONTACTS AND LOCATIONS:
Overall Officials: Mette Rosenkilde, MD, Study Director — University of Copenhagen
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No